CLINICAL TRIAL: NCT05024890
Title: WASH In Schools for Everyone (WISE): a Randomised Evaluation Assessing the Impact of a School-based Water, Sanitation and Hygiene (WASH) Intervention on Child Health and School Attendance in Addis Ababa, Ethiopia
Brief Title: The Impact of a School-based WASH Intervention on Child Health and School Attendance in Addis Ababa, Ethiopia
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Children's Investment Fund Foundation (Other); Splash (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17761
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2021-08

CONDITIONS: Diarrhea; Respiratory Tract Infections; Absenteeism
Keywords: water; sanitation; hygiene; schoolchildren; WASH in schools
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WASH in Schools programme (Experimental): Schools in the intervention group will receive the Splash WASH in Schools programme (Project WISE) during the study period (2021/2022 academic year), including sanitation, water storage and filtration, drinking water and handwashing stations, and hygiene and menstrual health education.
  Interventions: Other: Splash WASH in Schools programme (Project WISE)
- Control (No Intervention): Schools in the control group will receive no intervention during the study period (2021/2022 academic year), but will be on a waitlist to receive the Project WISE intervention after the end of the study period (2022/2023 academic year or later).

INTERVENTIONS:
Other: Splash WASH in Schools programme (Project WISE) — The Project WISE intervention includes:
  WASH infrastructure
  * Water storage tanks and water filtration systems
  * Durable plastic drinking water and handwashing stations
  * New/rehabilitated toilet facilities (gender-segregated, wheelchair-accessible, well-lit, ventilated, durable door and lock)
  Behaviour change promotion
  * Training of focal teachers to organise student 'hygiene club'
  * Annual soap drive and soap restocking
  * Behavioural 'nudges' (posters and mirrors at handwashing stations, colourful vests for hygiene clubs)
  MHM services
  * Toilets have water tap, bucket and waste bin
  * Emergency menstrual hygiene products available at school
  * Training of focal teachers to organise student 'gender club'
  * Education on puberty and menstruation for all pupils above 10 and parent resource guide
  Arms: WASH in Schools programme

SUMMARY:
This study aims to assess the effects of school-based, comprehensive water, sanitation, and hygiene improvements on child health and educational outcomes in schools in Addis Ababa, Ethiopia. Eligible schools will be randomly allocated to intervention or control groups. Data on pupil absence and illness will be collected longitudinally from students in selected classrooms in each school over the course of one academic year (2021/2022). This study will also assess the effects of the intervention on kindergarten students through parent interviews.

DETAILED DESCRIPTION:
This study uses a cluster-randomised controlled trial design to evaluate the impact of the WASH in Schools for Everyone (WISE) programme. Project WISE, implemented by Splash, aims to improve child health and attendance by 1) improving WASH infrastructure, 2) promoting WASH behaviour change and 3) strengthening menstrual hygiene management (MHM) services targeting girls aged 10 and above, in public schools across Addis Ababa.

60 public schools from planned implementation groups that will receive the WISE intervention will be randomised: 30 schools will be allocated to the intervention group (to receive the WISE intervention during the 2021/2022 academic year) and 30 schools will be allocated to the control group (on a waitlist to receive the WISE intervention after study completion). Randomisation will be stratified by school size (number of students) and presence of a kindergarten. In each selected school, between two and four classes will be randomly selected from grades 2-8 - to obtain a sample size of approximately 100 students in total per school. Students in the selected classes will be enrolled at the start of the academic year (September 2021) and followed up with unannounced visits every 4-6 weeks until the end of the academic year (May 2022). Primary outcomes of pupil-reported illness and absence will be assessed during enrolment and at each follow-up visit. Secondary outcomes are restricted to subsets of students by age and gender, and will be assessed during the final follow-up visit. Students joining the class mid-way through the year will be enrolled in the study, and students who leave the class will be recorded.

Key outcomes of interest are longitudinal prevalence of absence and illness (diarrhoea and respiratory infection) over the course of the academic year, measured as cumulative number of days absent/with illness per 100 school days after adjustment for child- and school-specific covariates. Data collected in intervention schools prior to and/or during the active Splash intervention will not be included in the primary impact evaluation analysis. Sub-population analysis of evaluation outcomes in girls post-menarche will allow assessment of the gendered effects of the intervention. We will also monitor intervention fidelity and compliance, as well as cost-effectiveness of the intervention, through routine data collection with students and school staff.

40 public schools with a kindergarten will be enrolled to assess the impacts of the intervention among kindergarten students (20 intervention, 20 control). Schools enrolled in the intervention and control arms of the main study among older children that have a kindergarten will be also enrolled in the kindergarten evaluation. If there are fewer than 20 such schools in each arm, additional kindergarten schools will be randomised (estimated 10 additional schools per arm). In each selected school, 20 kindergarten students will be randomly selected for participation. Parents of selected students will be invited to participate in weekly telephone surveys over a four-week period in February/March 2022 in order to assess the longitudinal prevalence of illness and absence among kindergarteners.

ELIGIBILITY:
Main study among older children (7-16 years)

School inclusion criteria:

* School is part of Splash Project WISE implementation groups
* School agrees to participate in the research

School exclusion criteria:

* School has received a water, sanitation, or hygiene intervention in the three years prior to study activities
* School is kindergarten only
* School is secondary only (grades 9 and above, equivalent)
* School provides education to vulnerable population groups only

Child inclusion criteria:

* Child is registered at a school that meets eligibility criteria and selected for the study
* Child is in grades 2-8
* Child's parents do not return the opt-out consent form
* Child provides assent to participate in the research

Child exclusion criteria:

* Child is unable to provide assent for data collection
* Child is 17 or older
* Child does not meet age eligibility for specific data collection activities

Kindergarten evaluation (4-6 years)

School inclusion criteria:

* School is part of Splash Project WISE implementation groups
* School has a kindergarten
* School agrees to participate in the research

School exclusion criteria:

* School has received a water, sanitation, or hygiene intervention in the three years prior to study activities
* School provides education to vulnerable population groups only

Child inclusion criteria:

* Child is registered at a school that meets eligibility criteria and selected for the study
* Child is in kindergarten
* Child's parent/guardian provides consent to participate in the research

Child exclusion criteria:

* Child is 7 or older

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7072 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Roll-call absence prevalence - Older children (7-16) | Longitudinal: Every 4-6 weeks. Participants will be followed for 9 months (September 2021-May 2022)
  Attendance on the day of data collection will be recorded for all children in selected classes. This indicator is collected longitudinally over the course of the study at follow-up visits every 4-6 weeks.
Self-reported absence prevalence - Older children (7-16) | Longitudinal: Baseline and every 4-6 weeks. Participants will be followed for 9 months (September 2021-May 2022)
  All children present in selected classes will be asked to report full- and partial-day absence over the past week of school. This indicator is collected longitudinally over the course of the study at follow-up visits every 4-6 weeks.
2- and 7-day period prevalence of diarrhoea - Older children (7-16) | Longitudinal: Baseline and every 4-6 weeks. Participants will be followed for 9 months (September 2021-May 2022)
  All children present in selected classes will be asked whether they have had diarrhoea within the past 2 and 7 days. This indicator is collected longitudinally over the course of the study at follow-up visits every 4-6 weeks.
2- and 7-day period prevalence of respiratory infection - Older children (7-16) | Longitudinal: Baseline and every 4-6 weeks. Participants will be followed for 9 months (September 2021-May 2022)
  All children present in selected classes will be asked whether they have had specific symptoms of respiratory infection within the past 2 and 7 days. This indicator is collected longitudinally over the course of the study at follow-up visits every 4-6 weeks.
Days with diarrhoea in past week - Kindergarten (4-6) | Longitudinal: Weekly for four weeks (February/March 2022).
  Parent-reported days with diarrhoea among kindergarten students with one-week recall period, assessed using telephone surveys. Cumulative days with diarrhoea over the four-week period will be calculated.
Days with respiratory infection in past week - Kindergarten (4-6) | Longitudinal: Weekly for four weeks (February/March 2022).
  Parent-reported days with symptoms of respiratory infection among kindergarten students with one-week recall period, assessed using telephone surveys. Cumulative days with respiratory infection over the four-week period will be calculated.
Absence in past week - Kindergarten (4-6) | Longitudinal: Weekly for four weeks (February/March 2022).
  Parent-reported days of absence from kindergarten with one-week recall period, assessed using telephone surveys. Cumulative absence over the four-week period will be calculated.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) total score - Older children (11-16) | Final follow-up at 9 months (May 2022)
  Children aged 11 or older in selected classrooms will complete the self-rated SDQ (25 items) as a measure of wellbeing.
Self-Efficacy in Addressing Menstrual Needs Scale (SAMN-Scale) total score - Older children (10-16) | Final follow-up at 9 months (May 2022)
  Post-menarcheal girls aged 10 or older present in selected classrooms will be asked to complete the SAMN-Scale questionnaire. SAMN-Scale measures respondents' perceived self-efficacy to address their menstrual needs.
Menstrual Practice Needs Scale (MPNS-36) total score - Older children (10-16) | Final follow-up at 9 months (May 2022)
  Post-menarcheal girls aged 10 or older present in selected classrooms will be asked to complete the MPNS-36 questionnaire. MPNS-36 measures the extent to which respondents' menstrual management practices and environments were perceived to meet their needs during their last period.

OTHER OUTCOMES:
Gender parity in school enrolment using the adjusted gender parity index (aGPI) | Baseline (September 2021) and end-of-year at 9 months (May 2022)
  School enrolment data will be collected at the start and end of the academic year to measure gender parity in enrolment.
Subjective wellbeing using smiley faces visual analogue scale - Older children (7-16) | Final follow-up at 9 months (May 2022)
  All children present in selected classrooms will be asked to rate their mood using a smiley faces visual analogue scale as a measure of subjective wellbeing.
Sanitation-related quality of life (SanQoL) total score - Older children (7-16) | Final follow-up at 9 months (May 2022)
  All children present in selected classrooms will complete the SanQoL questionnaire, a 5-item measure of sanitation-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreibelbis, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Oliver Cumming, MSc, Study Director — London School of Hygiene and Tropical Medicine; Elizabeth Allen, PhD, Study Director — London School of Hygiene and Tropical Medicine; Baptiste Leurent, PhD, Study Director — London School of Hygiene and Tropical Medicine; Sarah Bick, MSc, Study Director — London School of Hygiene and Tropical Medicine; Alem Ezezew, Study Director — Holster International Research & Development Consultancy
Locations (1):
- Holster International Research and Development Consultancy, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Bick S, Ezezew A, Opondo C, Leurent B, Argaw W, Hunter EC, Cumming O, Allen E, Dreibelbis R. Impact of a school-based water and hygiene intervention on child health and school attendance in Addis Ababa, Ethiopia: a cluster-randomised controlled trial. BMC Med. 2024 Sep 2;22(1):348. doi: 10.1186/s12916-024-03558-x. PMID 39218883